CLINICAL TRIAL: NCT01192425
Title: P06-001: (EX)Amination of (P)NH, by (L)Evel (O)f CD59 on (RE)d and White Blood Cells, in Bone Marrow Failure Syndromes
Brief Title: Paroxysmal Nocturnal Hemoglobinuria (PNH), Level of CD59 on Red and White Blood Cells in Bone Marrow Failure Syndromes
Acronym: EXPLORE
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Michael Bombara, Senior Director, Global Clinical Operations, Alexion Pharmaceuticals, Inc.
Other Study IDs: P06-001
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Hemoglobinuria
Keywords: PNH clone cells; Aplastic Anemia; AA; Myelodysplastic Syndromes; MDS; bone marrow failure syndromes; FLAER; Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria; Anemia, Aplastic; Myelodysplastic Syndromes; Bone Marrow Failure Disorders; Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Examine red and white blood cells of PNH patients with bone marrow failure syndromes.

ELIGIBILITY:
Inclusion Criteria:

* At least 10 years of age.
* Has aplastic anemia, myelodysplastic syndromes or other bone marrow failure syndromes

Exclusion Criteria:

* Has any condition that might interfere with the patient's participation

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at least 10 years of age with aplastic anemia, myelodyplastic syndromes or other bone marrow failure syndromes.
Sampling Method: Probability Sample
Enrollment: 5580 (Actual)